CLINICAL TRIAL: NCT03155828
Title: A Novel Method of Restoring Menstrual Cyclicity or Ovulatory Function in PCOS Patients: The Use of CPAP to Improve More Than Sleep Quality
Brief Title: Using CPAP to Improve Menstruation in Women With Polycystic Ovarian Syndrome and Obstructive Sleep Apnea
Status: Withdrawn | Type: Observational
Why Stopped: Lack of enrollment
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Kelly Pagidas, Professor, Obstetrics and Gynecology and Women's Health, University of Louisville
Other Study IDs: 16.0388
Record Dates: First submitted 2017-05-11; First posted 2017-05-16 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Sleep Apnea, Obstructive; Anovulation; Polycystic Ovarian Syndrome
Keywords: PCOS, OSA, CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive; Anovulation; Polycystic Ovary Syndrome; Microcephaly, Primary Autosomal Recessive, 6

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: CPAP — Women with diagnosed obstructive sleep apnea will be treated using continuous positive airway pressure as per standard of care.

SUMMARY:
The purpose of this study is to determine if treatment of obstructive sleep apnea (OSA) with continuous positive airway pressure in women with both OSA and polycystic ovarian syndrome will improve the regularity of the women's menstrual cycles.

DETAILED DESCRIPTION:
Women seeking fertility treatment at the University of Louisville will be screened for polycystic ovarian syndrome (PCOS) based on history and then blood work if history suggests PCOS. After establishing a diagnosis of PCOS based on the National Institute of Health criteria, they will be screened for impaired glucose tolerance, Class III obesity, and obstructive sleep apnea [using the Epworth Sleepiness Scale (ESS) as the initial screen]. For those women that screen positive on the ESS, they will be referred to the University of Louisville Physicians Sleep Center for a formal sleep study. Only patients with PCOS, severe obstructive sleep apnea, impaired glucose tolerance, and Class III obesity will qualify for enrollment in the study. Once enrolled, patients will be encouraged to use continuous positive airway pressure (CPAP, standard of care for treatment of obstructive sleep apnea) for at least six months. During those six months, patients will be asked to track their menstrual cycles and whether they took progesterone to induce a withdrawal bleed during that time period. The use of ovulation predictor kits to help determine ovulation status will be encouraged, but not required for the study.

During initial evaluation, patients seeking fertility care having a clinical presentation concerning for PCOS have their blood drawn for evaluation of thyroid stimulating hormone, free and total testosterone, antimullerian hormone, and 2 hour glucose tolerance test. At the conclusion of six months of CPAP therapy, patients will be asked to repeat the above blood tests for comparison to baseline values.

Women can continue to attempt pregnancy during the study time period if they desire.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35
* English speakers
* Polycystic ovarian syndrome by NIH criteria
* Abnormal 2 hour glucose tolerance test
* Body mass index >/= 40 kg/m2
* Severe obstructive sleep apnea diagnosed with either a home or in-house sleep study

Exclusion Criteria:

* Age <18 or >35
* Non English speakers
* No diagnosis of PCOS
* Normal glucose tolerance test
* No diagnosis of obstructive sleep apnea
* Body mass index < 40 kg/m2
* Using any form of hormonal contraception

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women seeking fertility treatment at the University of Louisville Reproductive Endocrinology and Infertility Center who have diagnosed polycystic ovarian syndrome, glucose intolerance, obesity, and obstructive sleep apnea.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Menstrual Cyclicity | 6 months
  Resumption of regular cycles as evaluated either by paper menstrual calendar or use of a menstrual cycle application on smart phone or tablet.

SECONDARY OUTCOMES:
Ovulation | 6 months
  Resumption of ovulatory cycles as evaluated by positive ovulation predictor kits.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Pagidas, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville Fertility Center, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No